CLINICAL TRIAL: NCT02692430
Title: LARGE SPONTANEOUS PORTOSYSTEMIC SHUNTS (SPSSs) IN PATIENTS WITH LIVER CIRRHOSIS. CLINICAL AND RADIOLOGICAL CHARACTERISTICS.
Brief Title: The International Imaging Registry in Liver Cirrhosis (BAVENO-VI SPSS GROUP).
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: IRCCS Policlinico S. Donato (Other); Martin-Luther-Universität Halle-Wittenberg (Other); Hospital Clinic of Barcelona (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Ramon y Cajal (Other); Odense University Hospital (Other); Puerta de Hierro University Hospital (Other); Royal Free Hospital NHS Foundation Trust (Other); University of Alberta (Other); University Hospital, Bonn (Other); University Hospital, Gasthuisberg (Other); Vienna General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LIVIMIAGE-129
Record Dates: First submitted 2016-02-10; First posted 2016-02-26 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2016-10

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Hepatic Encephalopathy
Keywords: Portosystemic Shunt; Hepatic encephalopathy; Portal hypertension; Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention is studied

SUMMARY:
The purpose of this study is to perform a multicentre registry of cirrhotic patients who had been submitted to an imagining technique in recent years (angio-CT scan or abdominal MRI), in order to collect anatomical and clinical information. The main objective will be focused on the study of portosystemic shunts and their relation with portal hypertension.

Patient with liver cirrhosis submitted to an abdominal angio-CT scan or a MRI from year 2010 to 2014 will be included in the study. The chosen imaging technique will be angio-CT preferably, but MRI data will also be available. Patients will be identified in every hospital by means of the registry of coded diagnoses and the lists of complementary tests performed. Clinical and radiological data of every patient will be collected. The clinical variables will be obtained from reviewing the patient clinical history. The radiological parameters will be gathered by means of the systematic review of the angio-CT or MRI.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* An evaluable imaging test (angio-CT or MRI) performed by any reason in the study period (from January 2010 to December 2014)

Exclusion Criteria:

* Presence of previous surgical shunts
* Prior liver transplant
* Neurological or psychiatric disorder that do not permit to establish the diagnosis of hepatic encephalopathy
* Presence of hepatocellular carcinoma beyond Milan criteria
* Terminal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients submitted to a angio-CT or MRI in several centres of international relevancy in the management of this condition.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of cirrhotic patients with a portosystemic shunt detected by angio-CT scan or MRI | 4 years
Number of cirrhotic patients that develop hepatic encephalopathy as a decompensation | 4 years

SECONDARY OUTCOMES:
Type of portosystemic shunts detected by angio-CT scan or MRI | 4 years
Number of cirrhotic patients that develop a decompensation (ascites, variceal bleeding, spontaneous bacterial peritonitis, hepatorenal syndrome) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan Genesca, MD, Principal Investigator — Vall d´Hebron Research Institut. Hospital Vall d´Hebron. Barcelona, Spain.
Locations (1):
- Vall d'Hebron Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Riggio O, Efrati C, Catalano C, Pediconi F, Mecarelli O, Accornero N, Nicolao F, Angeloni S, Masini A, Ridola L, Attili AF, Merli M. High prevalence of spontaneous portal-systemic shunts in persistent hepatic encephalopathy: a case-control study. Hepatology. 2005 Nov;42(5):1158-65. doi: 10.1002/hep.20905. PMID 16250033
- [Background] Laleman W, Simon-Talero M, Maleux G, Perez M, Ameloot K, Soriano G, Villalba J, Garcia-Pagan JC, Barrufet M, Jalan R, Brookes J, Thalassinos E, Burroughs AK, Cordoba J, Nevens F; EASL-CLIF-Consortium. Embolization of large spontaneous portosystemic shunts for refractory hepatic encephalopathy: a multicenter survey on safety and efficacy. Hepatology. 2013 Jun;57(6):2448-57. doi: 10.1002/hep.26314. Epub 2013 May 1. PMID 23401201
- [Background] Uflacker R, Silva Ade O, d'Albuquerque LA, Piske RL, Mourao GS. Chronic portosystemic encephalopathy: embolization of portosystemic shunts. Radiology. 1987 Dec;165(3):721-5. doi: 10.1148/radiology.165.3.3685350.
- [Background] Ohnishi K, Sato S, Saito M, Terabayashi H, Nakayama T, Saito M, Chin N, Iida S, Nomura F, Okuda K. Clinical and portal hemodynamic features in cirrhotic patients having a large spontaneous splenorenal and/or gastrorenal shunt. Am J Gastroenterol. 1986 Jun;81(6):450-5. PMID 3518409
- [Derived] Simon-Talero M, Roccarina D, Martinez J, Lampichler K, Baiges A, Low G, Llop E, Praktiknjo M, Maurer MH, Zipprich A, Triolo M, Vangrinsven G, Garcia-Martinez R, Dam A, Majumdar A, Picon C, Toth D, Darnell A, Abraldes JG, Lopez M, Kukuk G, Krag A, Banares R, Laleman W, La Mura V, Ripoll C, Berzigotti A, Trebicka J, Calleja JL, Tandon P, Hernandez-Gea V, Reiberger T, Albillos A, Tsochatzis EA, Augustin S, Genesca J; Baveno VI-SPSS group from the Baveno Cooperation. Association Between Portosystemic Shunts and Increased Complications and Mortality in Patients With Cirrhosis. Gastroenterology. 2018 May;154(6):1694-1705.e4. doi: 10.1053/j.gastro.2018.01.028. Epub 2018 Jan 31. PMID 29360462